CLINICAL TRIAL: NCT04060329
Title: Measuring and Improving Coproduction Using coopeRATE: A Before-and-after Study in Adult Cystic Fibrosis Care
Brief Title: Measuring and Improving Coproduction Using coopeRATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reasons associated with COVID-19 pandemic led to cancellation of Phase 2
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Glyn Jones-Elwyn, Professor, Trustees of Dartmouth College
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: SFD19152; ELWYN18QI0 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis; Chronic Disease
MeSH Terms: conditions — Cystic Fibrosis; Chronic Disease

STUDY DESIGN:
Intervention Model Description: In Phase 1, participants receive usual care only. In Phase 2, a different group of participants receive the coopeRATE Prompt intervention in addition to usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1 (No Intervention): Usual care
- Phase 2 (Experimental): Usual care + coopeRATE Prompt intervention
  Interventions: Behavioral: coopeRATE Prompt
- Clinicians (Other): After Phase 2, clinicians will be asked about their experiences with, and views about, the coopeRATE Prompt intervention.
  Interventions: Behavioral: coopeRATE Prompt

INTERVENTIONS:
Behavioral: coopeRATE Prompt — The coopeRATE Prompt intervention is a set of two questions delivered to patients immediately before the clinical encounter that elicit their concerns and goals.
  Arms: Clinicians; Phase 2

SUMMARY:
The purpose of this study is to identify new methods of measuring and improving collaborative goal setting between patients and clinicians in adult cystic fibrosis care.

DETAILED DESCRIPTION:
This study has 3 specific aims: Aim 1 will assess the construct validity of the coopeRATE Measure in the before phase of a before-and-after study in adult cystic fibrosis care settings. The coopeRATE Measure is a generic, patient-reported experience measure of collaborative goal setting that was recently developed in consultation with patients and other key stakeholders. Aim 2 will assess the impact of the coopeRATE Prompt intervention on collaborative goal setting and other outcomes in a before-and-after study in adult cystic fibrosis care settings. The coopeRATE Prompt intervention is a set of questions delivered to patients immediately before the clinical encounter that elicit their concerns and goals. Aim 3 will evaluate the feasibility and acceptability of implementing the coopeRATE Prompt and Measure in routine adult cystic fibrosis care.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of cystic fibrosis
2. Are 18 years of age or older
3. Can read and write in English
4. Are attending a participating site for a routine cystic fibrosis care visit
5. Have already consented to participate in the Cystic Fibrosis Foundation Patient Registry
6. Allow study researchers to access their Cystic Fibrosis Foundation Patient Registry information and link it to their study data
7. Have not previously participated in the study

Exclusion Criteria:

1. Do not have a diagnosis of cystic fibrosis
2. Are less than 18 years of age
3. Cannot read and write in English
4. Are not attending a participating site for a routine cystic fibrosis care visit
5. Have not already consented to participate in the Cystic Fibrosis Foundation Patient Registry
6. Do not allow study researchers to access their Cystic Fibrosis Foundation Patient Registry information and link it to their study data
7. Have previously participated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Collaborative goal setting | Immediately after the health care visit (Day 0)
  A new 3-item patient-reported measure under evaluation to assess collaborative goal setting between a patient and their clinician during the health care visit. Each item is rated on a 4-point scale ranging from 0 ('Strongly disagree') to 3 ('Strongly agree'), with an additional 'Not sure' option. Scoring method is to be determined.

SECONDARY OUTCOMES:
Shared decision-making | Immediately after the health care visit (Day 0)
  Patient-reported shared decision-making during the health care visit, assessed using the 3-item collaboRATE measure (Elwyn et al., 2013; Barr et al., 2014). Each item is rated on a 10-point scale ranging from 0 ('No effort was made') to 9 ('Every effort was made'). Respondent's are assigned a score of 1 if every item is rated 'Every effort was made' and a score of 0 for all other response combinations.
Interpersonal and communication skills | Immediately after the health care visit (Day 0)
  Patient-reported interpersonal and communication skills of their clinician during the health care visit, assessed using a 14-item version of the Communication Assessment Tool (CAT) (Makoul, Krupat, & Chang, 2007). Each item is rated on a 5-point scale ranging from 1 ('Poor') to 5 ('Excellent'). A respondent's total scale score is the percentage of items rated as 'Excellent'.
Self-efficacy to manage chronic disease | Immediately after the health care visit (Day 0)
  Patient-reported self-efficacy for managing their chronic disease immediately following the health care visit, assessed using an adapted version of the 6-item Self-Efficacy to Manage Chronic Disease Scale (Ritter & Lorig, 2014). Each item is rated on a 10-point scale ranging from 1 ('Not at all confident') to 10 ('Totally confident'). A respondent's total score is the mean of all item responses.

OTHER OUTCOMES:
Description of goals discussed during the visit | Immediately after the health care visit (Day 0)
  Patient-reported goals discussed during the health care visit (if goals were discussed), assessed using a single item with open-text response format.
Preference for discussing goals | Immediately after the health care visit (Day 0)
  Patient-reported preference for discussing goals with their clinician during the health care visit, assessed using a single item with multiple choice (single answer) format.
Use of coopeRATE Prompt | Immediately after the health care visit (Day 0) - Phase 2 only
  Patient-reported use of the coopeRATE Prompt intervention during the health care visit, assessed using a single item with multiple choice (single answer) format.
Reason(s) for not using coopeRATE Prompt (patient) | Immediately after the health care visit (Day 0) - Phase 2 only
  Patient-reported reason(s) for not using the coopeRATE Prompt intervention during the health care visit (if intervention was not used), assessed using a single item with multiple choice (multiple answer) format.
Perceived helpfulness of coopeRATE Prompt | Immediately after the health care visit (Day 0) - Phase 2 only
  Patient-reported perceived helpfulness of the coopeRATE Prompt intervention (if intervention was used), assessed using a single adapted item (Dalcin et al., 2015). The item is rated on a 5-point scale ranging from 0 ('Not at all helpful') to 4 ('Extremely helpful').
Way(s) in which coopeRATE Prompt helpful | Immediately after the health care visit (Day 0) - Phase 2 only
  Patient-reported way(s) in which the coopeRATE Prompt intervention was helpful (if intervention was perceived to be at least slightly helpful), assessed using a single item with multiple choice (multiple answer) format.
People seen during health care visit | Immediately after the health care visit (Day 0)
  Patient-reported people seen (e.g., doctor, nurse) during the health care visit, assessed using a single item with multiple choice (multiple answer) format.
History with people seen during health care visit | Immediately after the health care visit (Day 0)
  Patient-reported history with people seen during the health care visit, assessed using a single item with multiple choice (single answer) format.
Type of health care visit | Immediately after the health care visit (Day 0)
  Patient-reported type of health care visit, assessed using a single item with multiple choice (multiple answer) format.
Participation in other research | Immediately after the health care visit (Day 0)
  Patient-reported participation in other research studies during the health care visit, assessed using two single items with multiple choice (single answer) format.
Receipt of coopeRATE Prompt | Within one month after completion of Phase 2 patient data collection
  Clinician-reported receipt of the coopeRATE Prompt intervention, assessed using a single item with multiple choice (single answer) format.
Frequency of use of coopeRATE Prompt | Within one month after completion of Phase 2 patient data collection
  Clinician-reported frequency of using the coopeRATE Prompt intervention to guide conversations with patients (if intervention was ever received), assessed using a single item with multiple choice (single answer) format.
Reason(s) for not using coopeRATE Prompt (clinician) | Within one month after completion of Phase 2 patient data collection
  Clinician-reported reason(s) for not using the coopeRATE Prompt intervention to guide conversations with patients (if intervention was not always used), assessed using two single items with multiple choice (multiple answer) format.
Frequency of coopeRATE Prompt improving conversations | Within one month after completion of Phase 2 patient data collection
  Clinician-reported frequency of the coopeRATE Prompt intervention improving the quality of conversations with patients (if intervention was ever used), assessed using a single item with multiple choice (single answer) format.
Frequency of coopeRATE Prompt increasing consultation time | Within one month after completion of Phase 2 patient data collection
  Clinician-reported frequency of the coopeRATE Prompt intervention increasing consultation time with patients (if intervention was ever used), assessed using a single item with multiple choice (single answer) format.

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Elwyn, Principal Investigator — Dartmouth College
Locations (9):
- United States (9):
  - University of California San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center / Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center / Dartmouth-Hitchcock Manchester, Lebanon, New Hampshire
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elwyn G, Barr PJ, Grande SW, Thompson R, Walsh T, Ozanne EM. Developing CollaboRATE: a fast and frugal patient-reported measure of shared decision making in clinical encounters. Patient Educ Couns. 2013 Oct;93(1):102-7. doi: 10.1016/j.pec.2013.05.009. Epub 2013 Jun 12. PMID 23768763
- [Background] Barr PJ, Thompson R, Walsh T, Grande SW, Ozanne EM, Elwyn G. The psychometric properties of CollaboRATE: a fast and frugal patient-reported measure of the shared decision-making process. J Med Internet Res. 2014 Jan 3;16(1):e2. doi: 10.2196/jmir.3085. PMID 24389354
- [Background] Makoul G, Krupat E, Chang CH. Measuring patient views of physician communication skills: development and testing of the Communication Assessment Tool. Patient Educ Couns. 2007 Aug;67(3):333-42. doi: 10.1016/j.pec.2007.05.005. Epub 2007 Jun 18. PMID 17574367
- [Background] Ritter PL, Lorig K. The English and Spanish Self-Efficacy to Manage Chronic Disease Scale measures were validated using multiple studies. J Clin Epidemiol. 2014 Nov;67(11):1265-73. doi: 10.1016/j.jclinepi.2014.06.009. Epub 2014 Aug 3. PMID 25091546
- [Background] Dalcin AT, Jerome GJ, Fitzpatrick SL, Louis TA, Wang NY, Bennett WL, Durkin N, Clark JM, Daumit GL, Appel LJ, Coughlin JW. Perceived helpfulness of the individual components of a behavioural weight loss program: results from the Hopkins POWER Trial. Obes Sci Pract. 2015 Oct;1(1):23-32. doi: 10.1002/osp4.6. Epub 2015 Sep 9. PMID 27668085